CLINICAL TRIAL: NCT02400281
Title: Phase I-II Study of Crenolanib Combined With Standard Salvage Chemotherapy, and Crenolanib Combined With 5-Azacitidine in Acute Myeloid Leukemia Patients With FLT3 Activating Mutations
Brief Title: Study of Crenolanib Combined With Chemotherapy in FLT3-mutated Acute Myeloid Leukemia Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Arog Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARO-010
Record Dates: First submitted 2015-03-18; First posted 2015-03-27 (Estimated); Results first posted 2024-03-20 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Idarubicin; Cytarabine; Azacitidine; Mitoxantrone; Etoposide; etoposide phosphate; fludarabine; fludarabine phosphate; Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 crenolanib besylate combination (Experimental): Arm 1 patients will receive crenolanib besylate, combined with standard chemotherapy (Idarubicin/Cytarabine, MEC;Mitoxantrone/Etoposide/Cytarabine, FLAG-Ida: Fludarabine/Cytarabine/G-CSF/Idarubicin
  Interventions: Drug: Crenolanib besylate; Drug: Idarubicin; Drug: Cytarabine; Drug: Mitoxantrone; Drug: Etoposide; Drug: Fludarabine; Drug: G-CSF
- Arm 2 crenolanib besylate combination (Experimental): Arm 2 patients will receive crenolanib besylate and azacytidine.
  Interventions: Drug: Crenolanib besylate; Drug: Azacytidine

INTERVENTIONS:
Drug: Crenolanib besylate
  Other Names: CP-868,596-26
Drug: Idarubicin
  Other Names: 4-demethoxydaunorubicin
  Arms: Arm 1 crenolanib besylate combination
Drug: Cytarabine
  Other Names: cytosine arabinoside
  Arms: Arm 1 crenolanib besylate combination
Drug: Azacytidine
  Other Names: 5-azacytidine
  Arms: Arm 2 crenolanib besylate combination
Drug: Mitoxantrone
  Other Names: Novantrone
  Arms: Arm 1 crenolanib besylate combination
Drug: Etoposide
  Other Names: etoposide phosphate
  Arms: Arm 1 crenolanib besylate combination
Drug: Fludarabine
  Other Names: Fludarabine phosphate
  Arms: Arm 1 crenolanib besylate combination
Drug: G-CSF
  Arms: Arm 1 crenolanib besylate combination

SUMMARY:
This is an open label, two-arm, Phase I-II trial, non-randomized. Arm 1: crenolanib with standard chemotherapy (Idarubicin/Cytarabine, MEC;Mitoxantrone/Etoposide/Cytarabine, FLAG-Ida: Fludarabine/Cytarabine/G-CSF/Idarubicin) Arm 2: crenolanib with 5-azacitidine

DETAILED DESCRIPTION:
For each arm:

The phase I with dose-limiting toxicity (DLT) determination will use 3+3 design.

Phase II total of 52 patients (26 per arm) will be treated at established phase I dose.

Enrollment to be simultaneous to each arm.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed diagnosis of refractory/relapsed AML or high-risk MDS

   * Arm 1: Subjects must have received at least one prior therapy and a maximum of three prior therapies
   * Arm 2: Subjects must have received at least one prior therapy and a maximum of three prior therapies. No prior treatment with 5-Azacitidine is allowed in this arm.
2. FLT3 mutation positive (ITD, TKD or other)
3. ECOG PS 0-2
4. Adequate liver and renal function
5. Negative pregnancy test
6. Extramedullary leukemia allowed except CNS disease

Exclusion Criteria:

* Arm 1 and 2 Exclusion:

  1. <5% blasts in marrow or blood at time of screening
  2. Active HIV, hepatitis B or C
  3. CNS leukemia
  4. Clinically significant GVHD or organ dysfunction where chemotherapy specified by protocol cannot be given
  5. Patient with AML-M3 (APL)
  6. Pre-existing liver diseases (i.e. cirrhosis, chronic hepatitis B or C, nonalcoholic steatohepatitis, sclerosing cholangitis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2015-09; Primary Completion 2020-07-15 (Actual); Study Completion 2020-07-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Cortes, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Crenolanib With Standard Salvage Chemotherapy - Dose Level 1: Patients received 60 mg TID (dose level 1) crenolanib combined with standard salvage chemotherapy. Salvage chemotherapy options included IA (Idarubicin (Ida) 12 mg/m2 for 3 days (d) with cytarabine (AraC) 1.5 g/m2 for 4 days (3 d if age > 60 yrs)), FLAG-Ida (Fludarabine 30 mg/m2, AraC 2g/m2 each for 5 days, and Ida 8 mg/m2 for 3 days) or MEC (Mitoxantrone 8 mg/m2, etoposide 100 mg/m2, AraC 1g/m2 all for 5 days). Patients were allowed to continue receiving crenolanib for up to 365 days after the completion of cytotoxic therapy if they remained in remission. Standard rolling-6 design was implemented with dose escalation of crenolanib as follows: 60 mg TID (dose level 1), 80 mg TID (dose level 2), and 100 mg TID (dose level 3). Crenolanib was given continuously starting at the end of chemotherapy, and discontinued 3 days before the next cycle.
- Crenolanib With Standard Salvage Chemotherapy - Dose Level 2: Patients received 80 mg TID (dose level 2) crenolanib combined with standard salvage chemotherapy. Salvage chemotherapy options included IA (Idarubicin (Ida) 12 mg/m2 for 3 days (d) with cytarabine (AraC) 1.5 g/m2 for 4 days (3 d if age > 60 yrs)), FLAG-Ida (Fludarabine 30 mg/m2, AraC 2g/m2 each for 5 days, and Ida 8 mg/m2 for 3 days) or MEC (Mitoxantrone 8 mg/m2, etoposide 100 mg/m2, AraC 1g/m2 all for 5 days). Patients were allowed to continue receiving crenolanib for up to 365 days after the completion of cytotoxic therapy if they remained in remission. Standard rolling-6 design was implemented with dose escalation of crenolanib as follows: 60 mg TID (dose level 1), 80 mg TID (dose level 2), and 100 mg TID (dose level 3). Crenolanib was given continuously starting at the end of chemotherapy, and discontinued 3 days before the next cycle.
- Crenolanib With Standard Salvage Chemotherapy - Dose Level 3: Patients received 100 mg TID (dose level 3) crenolanib combined with standard salvage chemotherapy. Salvage chemotherapy options included IA (Idarubicin (Ida) 12 mg/m2 for 3 days (d) with cytarabine (AraC) 1.5 g/m2 for 4 days (3 d if age > 60 yrs)), FLAG-Ida (Fludarabine 30 mg/m2, AraC 2g/m2 each for 5 days, and Ida 8 mg/m2 for 3 days) or MEC (Mitoxantrone 8 mg/m2, etoposide 100 mg/m2, AraC 1g/m2 all for 5 days). Patients were allowed to continue receiving crenolanib for up to 365 days after the completion of cytotoxic therapy if they remained in remission. Standard rolling-6 design was implemented with dose escalation of crenolanib as follows: 60 mg TID (dose level 1), 80 mg TID (dose level 2), and 100 mg TID (dose level 3). Crenolanib was given continuously starting at the end of chemotherapy, and discontinued 3 days before the next cycle.
- Crenolanib With 5-azacitidine - Dose Level 1: Patients received 60 mg TID crenolanib combined with 5-azacitidine. 5-azacitidine was given at 75 mg/m2/day for 7 days each cycle. Patients were allowed to continue receiving crenolanib for up to 365 days after the completion of cytotoxic therapy if they remained in remission. Standard rolling-6 design was implemented with dose escalation of crenolanib as follows: 60 mg TID (dose level 1), 80 mg TID (dose level 2), and 100 mg TID (dose level 3). Crenolanib was given continuously starting at the end of chemotherapy, and discontinued 3 days before the next cycle.
- Crenolanib With 5-azacitidine - Dose Level 2: Patients received 80 mg TID crenolanib combined with 5-azacitidine. 5-azacitidine was given at 75 mg/m2/day for 7 days each cycle. Patients were allowed to continue receiving crenolanib for up to 365 days after the completion of cytotoxic therapy if they remained in remission. Standard rolling-6 design was implemented with dose escalation of crenolanib as follows: 60 mg TID (dose level 1), 80 mg TID (dose level 2), and 100 mg TID (dose level 3). Crenolanib was given continuously starting at the end of chemotherapy, and discontinued 3 days before the next cycle.
- Crenolanib With 5-azacitidine - Dose Level 3: Patients received 100 mg TID crenolanib combined with 5-azacitidine. 5-azacitidine was given at 75 mg/m2/day for 7 days each cycle. Patients were allowed to continue receiving crenolanib for up to 365 days after the completion of cytotoxic therapy if they remained in remission. Standard rolling-6 design was implemented with dose escalation of crenolanib as follows: 60 mg TID (dose level 1), 80 mg TID (dose level 2), and 100 mg TID (dose level 3). Crenolanib was given continuously starting at the end of chemotherapy, and discontinued 3 days before the next cycle.
Period: Overall Study
Arm/Group | Crenolanib With Standard Salvage Chemotherapy - Dose Level 1 | Crenolanib With Standard Salvage Chemotherapy - Dose Level 2 | Crenolanib With Standard Salvage Chemotherapy - Dose Level 3 | Crenolanib With 5-azacitidine - Dose Level 1 | Crenolanib With 5-azacitidine - Dose Level 2 | Crenolanib With 5-azacitidine - Dose Level 3
Started | 3 | 5 | 12 | 5 | 3 | 0
Completed | 3 | 5 | 10 | 5 | 2 | 0
Not Completed | 0 | 0 | 2 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Number of participants analyzed in the arm Crenolanib With 5-azacitidine - Dose Level 3 (100mg Crenolanib) is zero as the study concluded prior to enrolling any participants on this arm.
Groups:
- Total: Total of all reporting groups
Arm/Group | Crenolanib With Standard Salvage Chemotherapy - Dose Level 1 | Crenolanib With Standard Salvage Chemotherapy - Dose Level 2 | Crenolanib With Standard Salvage Chemotherapy - Dose Level 3 | Crenolanib With 5-azacitidine - Dose Level 1 | Crenolanib With 5-azacitidine - Dose Level 2 | Crenolanib With 5-azacitidine - Dose Level 3 | Total
Number analyzed (Participants) | 3 | 5 | 12 | 5 | 3 | 0 | 28
Age, Continuous [Median (Full Range); unit: years] | 43 [21 to 67] | 51 [30 to 58] | 65 [19 to 77] | 69 [37 to 81] | 60 [27 to 73] |  | 59.5 [19 to 81]
Age, Customized [Count of Participants; unit: Participants]
  18-60 years | 2 | 5 | 5 | 2 | 2 | 0 | 16
  >60 years | 1 | 0 | 7 | 3 | 1 | 0 | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 6 | 4 | 2 | 0 | 13
  Male | 2 | 5 | 6 | 1 | 1 | 0 | 15
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 1 | 0 | 1 | 0 | 0 | 0 | 2
  Asian | 0 | 0 | 1 | 0 | 0 | 0 | 1
  White | 2 | 4 | 7 | 4 | 2 | 0 | 19
  Other | 0 | 1 | 3 | 1 | 1 | 0 | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 3 | 1 | 0 | 0 | 5
  Not Hispanic or Latino | 3 | 4 | 8 | 3 | 3 | 0 | 21
  Unknown | 0 | 0 | 1 | 1 | 0 | 0 | 2
FLT3 Mutations [Count of Participants; unit: Participants] — Mutations in the gene encoding the trans-membrane tyrosine kinase FLT3. The type of FLT3 mutation detected by bone marrow assessment at diagnosis was collected. Subjects had either internal tandem duplications (ITD) in the juxtamembrane domain, point mutations or deletions in the tyrosine kinase domain (TKD) or both ITD and TKD mutations together.
  Participants
    ITD only | 1 | 1 | 3 | 2 | 3 | 0 | 10
    TKD only | 1 | 1 | 5 | 2 | 0 | 0 | 9
    ITD and TKD | 1 | 3 | 4 | 1 | 0 | 0 | 9
Baseline ECOG Performance [Count of Participants; unit: Participants] — ECOG performance status is graded by the investigator during a physical assessment. A greater ECOG grade is associated with greater impact of the disease on the ability of the subject to live. Grade 0 indicates subjects who are fully active and able to carry on all pre-disease performance. Grade 1 indicates subjects restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature. Grade 2 indicates subjects who are ambulatory and capable of all selfcare but unable to carry out any work activities.
  Participants
    0 | 1 | 1 | 1 | 1 | 0 | 0 | 4
    1 | 2 | 2 | 9 | 3 | 2 | 0 | 18
    2 | 0 | 2 | 2 | 1 | 1 | 0 | 6
Antecedent Hematological Disorder [Count of Participants; unit: Participants] — Whether or not subjects had a prior history of antecedent hematological disease. Subjects with de novo AML do not have a history of antecedent hematological disease, while subjects with secondary AML do.
  Participants | 0 | 3 | 4 | 3 | 0 |  | 10

OUTCOME MEASURES:

1. Primary Outcome: Response Rate of Crenolanib Besylate Combination Therapy
Description: To determine the response rate to crenolanib. CR Complete remission (CR) response criteria include a post-baseline bone marrow (BM) biopsy or aspiration % blasts <5%, absolute neutrophil count (ANC) >1×10^9/L and platelet count >100×10^9/L. CRi response included all CR criteria met, except participant did not experience either platelet recovery or ANC recovery. Morphologic Leukemia-Free State (MLFS) response included ≤5% in % blasts in the BM aspirate or biopsy. Resistant Disease (RD) was defined as the absence of CR, CRi, CRp, PR or MLFS. Death in aplasia response include deaths occurring following chemotherapy while cytopenic with an aplastic or hypoplastic BM prior to death without evidence of persistent leukemia.
Time Frame: Baseline up to first documented response, persistent disease, or death (whichever occurs first), 1 year.
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Crenolanib With Standard Salvage Chemotherapy - Dose Level 1 | Crenolanib With Standard Salvage Chemotherapy - Dose Level 2 | Crenolanib With Standard Salvage Chemotherapy - Dose Level 3 | Crenolanib With 5-azacitidine - Dose Level 1 | Crenolanib With 5-azacitidine - Dose Level 2 | Crenolanib With 5-azacitidine - Dose Level 3
Number analyzed (Participants) | 3 | 5 | 12 | 5 | 3 | 0
Participants
  CR/CRi | 2 | 0 | 3 | 1 | 1 | 0
  MLFS | 0 | 1 | 1 | 0 | 0 | 0
  ORR (CR/CRi+MLFS) | 2 | 1 | 4 | 1 | 1 | 0
  Persistent Disease (PD) | 1 | 3 | 7 | 4 | 2 | 0
  Death in Aplasia | 0 | 1 | 1 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From date of first dose up to 30-days after the last dose, 1 year.
Description: The number of participants at risk for Serious Adverse Events, All-Cause Mortality and Other Adverse Events is zero in the arm Crenolanib With 5-azacitidine - Dose Level 3 (100mg TID Crenolanib) as no patients were enrolled on this arm.
Arm/Group | Crenolanib With Standard Salvage Chemotherapy - Dose Level 1 | Crenolanib With Standard Salvage Chemotherapy - Dose Level 2 | Crenolanib With Standard Salvage Chemotherapy - Dose Level 3 | Crenolanib With 5-azacitidine - Dose Level 1 | Crenolanib With 5-azacitidine - Dose Level 2 | Crenolanib With 5-azacitidine - Dose Level 3
All-Cause Mortality (participants affected / at risk) | 3/3 | 5/5 | 8/12 | 5/5 | 3/3 | 0/0
Serious Adverse Events (participants affected / at risk) | 3/3 | 5/5 | 12/12 | 5/5 | 3/3 | 0/0
Other Adverse Events (participants affected / at risk) | 3/3 | 5/5 | 12/12 | 5/5 | 3/3 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Crenolanib With Standard Salvage Chemotherapy - Dose Level 1 (N=3) | Crenolanib With Standard Salvage Chemotherapy - Dose Level 2 (N=5) | Crenolanib With Standard Salvage Chemotherapy - Dose Level 3 (N=12) | Crenolanib With 5-azacitidine - Dose Level 1 (N=5) | Crenolanib With 5-azacitidine - Dose Level 2 (N=3) | Crenolanib With 5-azacitidine - Dose Level 3 (N=0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 3 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Melaena (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Catheter site haemorrhage (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Bacteraemia (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Lung infection (Infections and infestations) | 0 | 0 | 2 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 1 | 0 | 1 | 0 | 0
Pneumonia fungal (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0
Pseudomonas infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0
Septic arthritis staphylococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 2 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Crenolanib With Standard Salvage Chemotherapy - Dose Level 1 (N=3) | Crenolanib With Standard Salvage Chemotherapy - Dose Level 2 (N=5) | Crenolanib With Standard Salvage Chemotherapy - Dose Level 3 (N=12) | Crenolanib With 5-azacitidine - Dose Level 1 (N=5) | Crenolanib With 5-azacitidine - Dose Level 2 (N=3) | Crenolanib With 5-azacitidine - Dose Level 3 (N=0)
Anemia (Blood and lymphatic system disorders) | 3 | 5 | 9 | 5 | 2 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 3 | 2 | 5 | 0 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1 | 3 | 1 | 0 | 0
Splenomegaly (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 3 | 2 | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 1 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 1 | 1 | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 4 | 2 | 1 | 0 | 0
Arnold-Chiari malformation (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0 | 0 | 0
Ear discomfort (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 2 | 0 | 0 | 0
Otorrhoea (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0
Conjunctival oedema (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 2 | 1 | 1 | 0
Erythema of eyelid (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0
Eye pain (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0
Eye pruritus (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0
Lacrimation increased (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0
Ocular hyperaemia (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0
Periorbital oedema (Eye disorders) | 1 | 0 | 1 | 0 | 1 | 0
Photophobia (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 1 | 1 | 1 | 0 | 0
Vision impaired (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 2 | 0 | 4 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Anal fissure (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 1 | 5 | 4 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 2 | 9 | 2 | 2 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 2 | 1 | 0 | 0
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 1 | 2 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 | 1 | 2 | 0 | 1 | 0
Gingival recession (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Gingival swelling (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Lip pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Melaena (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 1 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 3 | 4 | 6 | 3 | 3 | 0
Odonophagia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Oral mucosal blistering (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 4 | 4 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 4 | 4 | 0 | 0
Asthenia (General disorders) | 0 | 1 | 1 | 0 | 0 | 0
Catheter site erythema (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Catheter site pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Catheter site haemorrhage (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Chills (General disorders) | 2 | 4 | 4 | 0 | 0 | 0
Face oedema (General disorders) | 0 | 1 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 1 | 4 | 7 | 3 | 2 | 0
Gait disturbance (General disorders) | 1 | 0 | 2 | 0 | 0 | 0
Generalised oedema (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Local swelling (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Localised oedema (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 2 | 1 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 2 | 1 | 1 | 0 | 0
Oedema peripheral (General disorders) | 2 | 3 | 5 | 1 | 2 | 0
Pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 5 | 4 | 2 | 0 | 0
Anorectal cellulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 2 | 2 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Abscess limb (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Burkholderia infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 1 | 1 | 0 | 0 | 0
Clostridium colitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 2 | 2 | 0 | 0 | 0
Candida infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Escherichia bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Lung infection (Infections and infestations) | 0 | 0 | 2 | 0 | 1 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 2 | 1 | 1 | 1 | 0 | 0
Pneumonia fungal (Infections and infestations) | 0 | 3 | 1 | 1 | 0 | 0
Pneumonia bacterial (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0
Pneumonia viral (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Pseudomonal bacteraemia (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0
Pseudomonas infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Rash pustular (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 1 | 1 | 1 | 0 | 0
Septic arthritis staphylococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Staphylococcal bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Septic shock (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Trichosporon infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0
Urinary tract infection enterococcal (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Viral sinusitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Eye injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1 | 0
Subdural hemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Transfusion reaction (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 2 | 3 | 4 | 3 | 2 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 2 | 3 | 1 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 3 | 2 | 3 | 3 | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 4 | 2 | 2 | 1 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 3 | 0 | 0 | 0
Blood creatinine decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
International normalised ratio increased (Investigations) | 1 | 1 | 0 | 0 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Blood urea increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Platelet count decreased (Investigations) | 1 | 2 | 3 | 3 | 1 | 0
Weight decreased (Investigations) | 0 | 1 | 1 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 2 | 1 | 2 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 4 | 4 | 1 | 0
Fluid overload (Metabolism and nutrition disorders) | 1 | 0 | 2 | 1 | 0 | 0
Fluid retention (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 4 | 7 | 3 | 2 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 2 | 2 | 0 | 0 | 0
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 3 | 4 | 3 | 0 | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 2 | 1 | 0
Hypoalbunaemia (Metabolism and nutrition disorders) | 3 | 5 | 8 | 4 | 2 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 3 | 5 | 7 | 3 | 2 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 4 | 7 | 4 | 2 | 0
Hypomagnaesemia (Metabolism and nutrition disorders) | 3 | 4 | 8 | 4 | 2 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 5 | 5 | 3 | 2 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 2 | 4 | 3 | 1 | 1 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hypouricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 3 | 2 | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 3 | 0 | 2 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2 | 0 | 1 | 0
Carcinoma in situ of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 1 | 3 | 0 | 2 | 0
Dysguesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Haemorrhage inctracranial (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 3 | 1 | 4 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 2 | 1 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Restless legs syndrome (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 2 | 2 | 2 | 0
Confusional state (Psychiatric disorders) | 1 | 0 | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 4 | 1 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 1 | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 1 | 0 | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 1 | 1 | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 9 | 3 | 2 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 4 | 3 | 2 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 3 | 1 | 2 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 2 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 1 | 1 | 0
Nasal crusting (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 0 | 2 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 2 | 0 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pneumonia respiratory synctial viral (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 2 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 1 | 1 | 0
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Endodontic procedure (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 0 | 0
Micrographic skin surgery (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 2 | 1 | 2 | 0
Hypotension (Vascular disorders) | 2 | 2 | 3 | 2 | 1 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pallor (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-05-18): https://cdn.clinicaltrials.gov/large-docs/81/NCT02400281/Prot_SAP_000.pdf